CLINICAL TRIAL: NCT05382637
Title: Growth Hormone in a Patient With a Dominant-Negative GHR Mutation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Andrew Dauber, Chief of Endocrinology, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000211
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Growth Disorders
MeSH Terms: conditions — Growth Disorders | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Growth hormone (Experimental): The participant will receive escalating dose of growth hormone until an IGF-1 level is maintained between the mean and +2 standard deviations.
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Daily growth hormone at a starting dose of 50 mcg/kg/day and escalating

SUMMARY:
This is a prospective interventional study designed for a single patient with a dominant-negative mutation in the growth hormone receptor gene (GHR) which results in increased levels of growth hormone binding protein (GHBP). The patient will receive escalating doses of growth hormone titrated to achieve an insulin like growth factor-1 level above the mean and then growth response to therapy will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Be the specific subject with the a specific mutation in GHR leading to high GHBP.

Exclusion Criteria:

There are no exclusion criteria for this study.

Min Age: 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2028-09-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Dauber, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Growth Hormone
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 1
Arm/Group | Growth Hormone
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 9.75 [9.75 to 9.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
Baseline Height standard deviation score [Number; unit: Standard deviation score from the CDC] — Baseline height standard deviation score based on the US CDC growth chart data. The CDC provides tables of both height percentiles and standard deviations of the distribution of heights by age and sex. The CDC has a SAS program that allows for calculation of an individual's height standard deviation score based on the population data. This is the standard way that height is recorded in many growth studies.
  Standard deviation score from the CDC | -3.18

OUTCOME MEASURES:

1. Primary Outcome: Growth Hormone Dose
Description: Dose of growth hormone required in mg/kg/day to achieve an IGF-1 level above the mean
Time Frame: 1 year
Measure: Number; unit: mg/kg/day
Arm/Group | Growth Hormone
Number analyzed (Participants) | 1
mg/kg/day | 0.250

2. Secondary Outcome: Growth Velocity
Description: Growth velocity during 1st year of growth hormone treatment
Time Frame: 1 year
Measure: Number; unit: cm/year
Arm/Group | Growth Hormone
Number analyzed (Participants) | 1
cm/year | 8.7

3. Secondary Outcome: Height Standard Deviation Score Using Center for Disease Control (CDC) Growth Chart
Description: Change in age and sex adjusted height standard deviation score based on the US CDC growth charts over the course of the 1st year of treatment with growth hormone. Height standard deviation score based on the US CDC growth chart data. The CDC provides tables of both height percentiles and standard deviations of the distribution of heights by age and sex. The CDC has a SAS program that allows for calculation of an individual's height standard deviation score based on the population data. This is the standard way that height is recorded in many growth studies.
Time Frame: Baseline to 1 Year
Measure: Number; unit: Standard deviations
Arm/Group | Growth Hormone
Number analyzed (Participants) | 1
Standard deviations | 0.81

ADVERSE EVENTS:
Time Frame: 1 year of study
Arm/Group | Growth Hormone
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT05382637/Prot_SAP_000.pdf